CLINICAL TRIAL: NCT06035289
Title: Klinisches Register Schweres Asthma
Brief Title: Register Schweres Asthma - German Asthma Net e.V.
Status: Recruiting | Type: Observational
Sponsor: German Asthma Net e.V. (Other)
Collaborators: AstraZeneca (Industry); GlaxoSmithKline (Industry); Sanofi (Industry); Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2018-13614
Record Dates: First submitted 2023-07-25; First posted 2023-09-13 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-10

CONDITIONS: Severe Asthma
Keywords: Registry; Biological
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The German Asthma Net e.V. focusses on science and research in patients with severe asthma. This includes, in particular, the optimization of medical care and treatment for patients with severe asthma as well as the elucidation and information. An unavoidable basis for a better understanding of severe asthma is the registration and comprehensive characterization of a large patient population. To date, there are only few reliable data on incidence, prevalence, phenotypes and treatment of patients with severe asthma. For this reason, the German Asthma Net e.V. was established in December 2011 as a clinical registry for patients with severe asthma, initially set up on a national basis.

DETAILED DESCRIPTION:
Sociodemographic parameters (e.g., gender, date of birth) and medical parameters (diagnosis, therapy) are entered in the register. In addition, data on lung function, laboratory values (IgE and eosinophil granulocytes), asthma control (symptoms, nocturnal awakenings, on-demand medication, exacerbations), smoking status, and concomitant therapy (inhalable corticosteroids, bronchodilators, and systemic steroids) are collected. This information will be collected at the baseline visit, and then once a year at a follow up visit, for fifteen years.

Participants will be assigned a unique study ID to protect the confidentiality of their personal health care information. Personal data and register data are on separate servers and thus meet the requirements of data protection.

The primary purpose is to establish a clinical registry for patients with severe asthma. The number of patients with severe asthma at a single center or practice is usually small, so several centers (clinics and practices) in Germany have joined together to form the German Asthma Net e.V. to optimize the diagnostic evaluation and treatment of patients with severe asthma.

ELIGIBILITY:
Definition: Severe asthma in children and adolescents

Poor symptom control in the last year despite (medium to) high doses of anti-inflammatory maintenance treatment:

(i) Age 6-18 years (at inclusion) (ii) Asthma diagnosis made by a medical doctor (iii) Potential differential diagnoses excluded (iv) Good compliance and trained inhalation technique (v) Evidence of:

a. Positive bronchodilator reversibility testing (≥ 12% increase in FEV1 after SABA) or b. Significant bronchial hyperreactivity (BHR) after unspecific provocation test (e.g. methacholine challenge or treadmill) according to ATS criteria (Am J Respir Crit Care Med 2000) (vi) High level of treatment:

1. Maintenance treatment with high doses of ICS (>400 μg budesonide or equivalent / ≥ 200 μg of fluticasone as monotherapy) or
2. Maintenance treatment with medium to high doses of ICS (≥400 μg budesonide or equivalent / ≥ 200 μg fluticasone) combined with LABA and/or LTRA and/or theophylline or
3. Treatment with oral steroids for ≥ 3 months (vii) Poor asthma control:

a. Inadequate symptom in the past 4 weeks: i. asthma symptoms ≥3 x / week or use of rescue medication ≥3 x / week; or ii. activity limitations due to asthma; or iii. any nighttime asthma symptoms; or b. ≥ 1 exacerbation in the last year with ≥ 3 days of OCS treatment or hospitalisation or b. Poor lung function with reduced Tiffeneau index or FEV1 at inclusion (viii) written informed consent (parent or legal guardian)

Exclusion criteria:

(i) Diagnosis of other obstructive or systemic pulmonary diseases (e.g. cystic fibrosis, COPD) despite BPD at inclusion (ii) Other congenital lung diseases or pulmonary malformations (iii) Other significant chronic diseases (iv) Congenital or acquired heart defects with significant functional limitations

Definition: Severe asthma in adults

High level of treatment (A), i.e. step 5 of GINA guideline or (B) medium level of treatment and poor symptom control:

(A) High level of treatment:

1. Maintenance treatment with high-dose inhaled corticosteroids (≥ 1000 μg beclomethasone (BDP, powder) or equivalent) in combination with LABA or LTRA or theophylline or
2. Maintenance treatment with oral corticosteroids (OCS) for ≥3 months independent of other asthma treatments or
3. Treatment with monoclonal antibodies independent of other asthma treatments

B) Medium level of treatment and poor symptom control:

1. Maintenance treatment with medium to high doses of ICS (≥ 500 μg BDP (powder) or equivalent) in combination with LABA or LTRA or theophylline and
2. Poor symptom control:

(i) asthma symptoms ≥ 3 x / week or use of rescue medication ≥ 3 x / week; or (ii) activities limited due to asthma; or (iii) any nighttime asthma symptoms; or (iv) ≥ 1 exacerbation in the last year with ≥ 3 days of OCS treatment or (v) FEV1<80% of predicted

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients presenting to participating study center (pulmonologists in private practice or in pulmonary departments in hospital)
Sampling Method: Non-Probability Sample
Enrollment: 4500 (Estimated)
Dates: Start 2011-11-01 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Symptom Control | Baseline, four months, yearly for up to 15 years
  Changes in symptom control at baseline and during the follow-up period and at study end using the Asthma Control Test (ACT).

SECONDARY OUTCOMES:
Exacerbations | Baseline, four months, yearly for up to 15 years
  Number of exacerbation with/without hospitalization
Utilization of the health care system | Baseline, yearly for up to 15 years
  Number of visits at a pneumologist/ specialist, number of emergency consultations, number of hospitalizations, number of rehabilitation stays
Symptoms and health-related quality of life | Baseline, yearly for up to 15 years
  Asthma Control Test (ACT: 5 questions, scale 1- 5, min score 5, max score 25, the lower the score the better the Asthma control)
Quality of Life Questionnaire | Baseline, yearly for up to 15 years
  Mini Asthma Quality of Life Questionnaire (Mini-AQLQ: 15 questions, scale 1 to 7, min score 15, max score 105, the higher the score, the better the quality of life)
Asthma Control Questionnaire | Baseline, yearly for up to 15 years
  Asthma Control Questionnaire ACQ: 5 questions, scale 0 to 6, min score 0, max score 30, the lower the score the better the Asthma control)
Forced Exhaled Volume in 1 second (FEV1) | Baseline, 4 months, yearly for up to 15 years
  FEV1 at consultation, FEV1 last 2 years, changes in FEV1 in liter from the target value
Forced Vital Capacity (FVC) | Baseline, 4 months, yearly for up to 15 years
  FVC at consultation, FEV1 last 2 years, changes in FEV1 in liter from the target value
Changes in medication | Baseline, 4 months, yearly for up to 15 years
  changes in substances if there is a new drug used.
Changes in dose in mg | 4 months, yearly for up to 15 years
  Changes in dose in mg
Fraction of exhaled nitric oxide (FeNo) | Baseline, 4 months, yearly for up to 15 years
  Changes in FeNo in ppb
Blood Gas analysis | Baseline, 4 months, yearly for up to 15 years
  pO2 in kPa/ mmHg, pCO2 in kPa/ mmHg
Blood Gas analysis | Baseline, 4 months, yearly for up to 15 years
  Blood-oxygen saturation in %
Leucocytes | Baseline, 4 months, yearly for up to 15 years
  Changes in leucocytes in nl
Neutrophilic granulocytes | Baseline, 4 months, yearly for up to 15 years
  Changes in Neutrophilic granulocytes in nl or %
Eosinophilic granulocytes | Baseline, 4 months, yearly for up to 15 years
  Changes in Eosinophilic granulocytes in µl or %
CO diffusion capacity | Baseline, yearly for up to 15 years
  Changes in mmol/min/kPa/ %

CONTACTS AND LOCATIONS:
Locations (45):
- Germany (45):
  - Kardiologische und fachinternistische ÜBAG Dr. Sandrock und Partner, Altdorf
  - Universitätsklinikum Augsburg Kinderpulmologie und -allergologie, Augsburg
  - Praxis Dr. Grün, Bad Windsheim
  - CIMS Studienzentrum Bamberg, Bamberg
  - Lungenpraxis Tegel, Berlin
  - Evangelisches Klinikum Bethel v. Bodelschwinghsche Stiftungen Bethel, Bielefeld
  - Helios Lungen- und Allergiezentrum Bonn, Bonn
  - Universitätsnedizin Bonn, Bonn
  - Zentrum für Kinderheilkunde, Klinik und Poliklinik für Allgemeine Pädiatrie, Allergieabteilung, Bonn
  - Lungenpraxis Medicum Böblingen, Böblingen
  - Prof.-Hess-Kinderklinik Bremen-Mitte, Bremen
  - MECS Cottbus, Cottbus
  - Evangelisches Krankenhaus Düsseldorf, Düsseldorf
  - Lunge im Zentrum, Erlangen
  - Universitätsmedizin Essen, Essen
  - Pneumologie am Schelztor Esslingen, Esslingen am Neckar
  - Praxis Dr. Herden, Freising
  - ALB FILS Kliniken, Göppingen
  - Hamburger Institut für Therapieforschung GmbH, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Praxisgmeinschaft Dr. Abenhardt und Jochen Hinrichs-Pavlik, Heidelberg
  - Thoraxklinik Heidelberg gGmbH, Heidelberg
  - Lungenarztpraxis Dr. Hubatsch, Heilbronn
  - Atemwegszentrum Kaiserslautern, Kaiserslautern
  - MVZ Klinikum Kempten, Kempten
  - Pneumologische Gemeinschaftspraxis, Koblenz
  - Lungenpraxis Konstanz, Konstanz
  - DONAUISAR Klinikum Deggendorf-Dingolfing-Landau, Landau an der Isar
  - Asthma Allergiezentrum, Leverkusen
  - Lungenfachklinik Medizinische Klinik I, Pneumologie, Löwenstein
  - IKF Pneumologie GmbH & Co. KG, Mainz
  - Lungenfacharztpraxis Dr. C. Lüttecke-Hecht, Mainz
  - Lungenfacharztpraxis Dr. Gall, Mainz
  - Univsersitätsmedizin Mainz, Mainz
  - Dr. von Haunersches Kinderspital, München
  - LMU Klinikum der Universität München, Ambulanz für Schweres Asthma (Erwachsene), München
  - Universitätsklinikum Regensburg, Regensburg
  - Universitätsmedizin Rostock, Med. Klinik I, Abt. Pneumologie & Interdiszipl. Internistische Intensivmedizin, Rostock
  - Lungenpraxis Schleswig/ Respiratio, Schleswig
  - Ambulante Pneumologie mit Allergiezentrum (BAG), Stuttgart
  - RBK Lungenzentrum Stuttgart, Stuttgart
  - Internistische Gemeinschaftspraxis Bitburg-Trier, Trier
  - Uniklinik Ulm, Sektion Pneumologie, Klinik für Innere Medizin II, Ulm
  - Fachkliniken Wangen, Wangen
  - Marien-Hospital, Klinik für Kinder- und Jugendmedizin, Wesel

REFERENCES:
- [Result] Bal C, Pohl W, Milger K, Skowasch D, Schulz C, Gappa M, Koerner-Rettberg C, Jandl M, Schmidt O, Zehetmayer S, Taube C, Hamelmann E, Buhl R, Korn S, Idzko M; German Asthma Net (GAN) study group. Characterization of Obesity in Severe Asthma in the German Asthma Net. J Allergy Clin Immunol Pract. 2023 Nov;11(11):3417-3424.e3. doi: 10.1016/j.jaip.2023.06.049. Epub 2023 Jul 4. PMID 37406803
- [Result] Milger K, Suhling H, Skowasch D, Holtdirk A, Kneidinger N, Behr J, Timmermann H, Schulz C, Schmidt O, Ehmann R, Hamelmann E, Idzko M, Taube C, Lommatzsch M, Buhl R, Korn S. Response to Biologics and Clinical Remission in the Adult German Asthma Net Severe Asthma Registry Cohort. J Allergy Clin Immunol Pract. 2023 Sep;11(9):2701-2712.e2. doi: 10.1016/j.jaip.2023.05.047. Epub 2023 Jun 8. PMID 37301433
- [Result] Korn S, Milger K, Skowasch D, Schulz C, Mohrlang C, Wernitz M, Paulsson T, Hennig M, Buhl R. Real-World Experience on the Use of Mepolizumab from the Severe Asthma Registry of the German Asthma Net (MepoGAN-Study). J Asthma Allergy. 2023 May 11;16:541-552. doi: 10.2147/JAA.S403286. eCollection 2023. PMID 37197193
- [Result] Milger K, Skowasch D, Hamelmann E, Mummler C, Idzko M, Gappa M, Jandl M, Korner-Rettberg C, Ehmann R, Schmidt O, Taube C, Holtdirk A, Timmermann H, Buhl R, Korn S. Bronchodilator Reversibility in the GAN Severe Asthma Cohort. J Investig Allergol Clin Immunol. 2023 Dec 14;33(6):446-456. doi: 10.18176/jiaci.0850. Epub 2022 Aug 24. PMID 36000830
- [Result] Bal C, Idzko M, Skrgat S, Koch A, Milger K, Schulz C, Zehetmayer S, Hamelmann E, Buhl R, Korn S; collaborators from the German Asthma Net (GAN). Fraction of exhaled nitric oxide is associated with disease burden in the German Asthma Net severe asthma cohort. Eur Respir J. 2022 Jun 2;59(6):2101233. doi: 10.1183/13993003.01233-2021. Print 2022 Jun. PMID 35273030
- See also: Website — http://www.germanasthmanet.de